CLINICAL TRIAL: NCT07143357
Title: Development of a Dyadic Mind-body Program for Cardiac Arrest Survivors and Their Caregivers: Recovering Together After Cardiac Arrest (RT-CA).
Brief Title: Mind-body Resilience Program for Cardiac Arrest Survivors and Their Caregivers: Recovering Together After Cardiac Arrest
Acronym: RT-CA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Alexander Presciutti, Member of the Faculty, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P002063; 5K23AT012487 (NIH)
Record Dates: First submitted 2025-08-05; First posted 2025-08-27 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Emotional Distress; Cardiac Arrest (CA); Anxiety; Depression; Caregivers; Survivorship; Resilience; Mindfulness
Keywords: emotional distress; cardiac arrest; cardiac arrest survivorship; caregivers; resilience; mindfulness; mind-body; behavioral interventions; anxiety; depression
MeSH Terms: conditions — Heart Arrest; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovering Together after Cardiac Arrest 1 (Experimental): Dyads will participate in 6 30-minute skills-based sessions. Sessions will also include provision of anticipatory guidance and and resources to manage cardiac arrest-specific stressors. A clinical psychologist will deliver all of the sessions. The main intervention goal is to provide dyads with resiliency skills and resources to reduce emotional distress and prevent chronic distress.
  Interventions: Behavioral: Recovering Together after Cardiac Arrest 1
- Recovering Together after Cardiac Arrest 2 (Other): Recovering Together after Cardiac Arrest is a minimally enhanced usual care control. Dyads will participate in one 30-minute session with a clinician reviewing available psychosocial resources for cardiac arrest survivors and their caregivers.
  Interventions: Other: Recovering Together after Cardiac Arrest 2

INTERVENTIONS:
Behavioral: Recovering Together after Cardiac Arrest 1 — The intervention will teach resiliency skills (mindfulness and coping) to dyads and provider anticipatory guidance and resources to manage stressors specific to cardiac arrest. These sessions will take place in person until the survivor is discharged; remaining sessions will occur over Zoom.
  Arms: Recovering Together after Cardiac Arrest 1
Other: Recovering Together after Cardiac Arrest 2 — In this minimally enhanced usual care control, dyads will participate in one 30-minute session with a clinician at beside to review a pamphlet of available psychosocial resources for cardiac arrest survivors and their caregivers.
  Arms: Recovering Together after Cardiac Arrest 2

SUMMARY:
The purpose of this study is to pilot two resilience interventions for cardiac arrest survivors and their informal caregivers, Recovering Together after Cardiac Arrest 1 and Recovering Together after Cardiac Arrest 2 . The data the investigators gather in this study will be used to further refine the interventions.

DETAILED DESCRIPTION:
The goal of this study is to test the feasibility of our proposed interventions through a pilot RCT. The investigators will deliver the RCT intervention (N=42 dyads; 84 participants total) and evaluate feasibility and acceptability based on a priori benchmarks.

The RCT will initially take place at Massachusetts General Hospital intensive care units and step-down units. Cardiac arrest survivor-caregiver dyads will be randomly assigned to one of two groups - Recovering Together after Cardiac Arrest 1 (RT-CA 1) or Recovering Together after Cardiac Arrest 2 (RT-CA 2).

RT-CA 1 involves six, 30-minute weekly sessions beginning at bedside and continuing over Zoom after the survivor is discharged. RT-CA 2 involves one, 30 minute session at bedside.

All participants will complete psychosocial survey measures at baseline, six weeks, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Out-of-hospital or in-hospital CA survivor (must have new diagnosis of "cardiac arrest" in electronic medical record from index hospitalization with documented loss of pulse) with an identified caregiver (identified by the survivor who is their primary source of emotional and functional support)
2. survivor must score >5 on Short Form of the Mini Mental State Exam for sufficient cognitive function for meaningful participation
3. ability and willingness to participate in a hybrid in-person/live video intervention
4. English speaking adults (18 year or older)
5. at least one member of the dyad endorses clinically significant emotional distress during screening (>7 on either of the Hospital Anxiety and Depression Scale subscales).

Exclusion Criteria:

1. active psychosis, mania, substance dependence, or suicidal intent or plan that would require a higher level of care
2. any other psychiatric or neurological condition that would preclude meaningful participation
3. the caregiver must not be a cardiac arrest survivor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment | pre-test
  Proportion of eligible dyads that consent to participation
Feasibility of Randomization | The end of treatment at 6 weeks
  Proportion of randomized participants who submit post-test assessments
Feasibility of Assessment Completion | pre-test, the end of treatment at 6 weeks, and 3 months after the end of treatment
  Proportion of participants with no assessment measures missing at pre-test, post-test, and 3 month follow-up
Feasibility of Program Adherence (RT-CA 1) | the end of treatment at 6 weeks
  Proportion of RT-CA 1 dyads that initiate the program by attending session 1 and complete at least 4 of 6 sessions.
Therapist Fidelity | the end of treatment at 6 weeks
  Proportion of 20% randomly-selected RT-CA 1 sessions in which the therapist fully adheres to program content, ascertained by a fidelity checklist
Treatment Satisfaction (RT-CA 1) | the end of treatment at 6 weeks
  Proportion of RT-CA 1 participants that endorse satisfaction, defined as above the midpoint on the Client Satisfaction Questionnaire-3
Credibility (RT-CA 1) | pre-test
  Proportion of RT-CA 1 participants that endorse program credibility at pre-test, defined as scoring above the midpoint on the Credibility sub scale of the Credibility/Expectancy Questionnaire
Expectancy (RT-CA 1) | pre-test
  Proportion of RT-CA 1 participants that endorse expectancy to improve. from the program at pre-test, defined as scoring above the midpoint on the Expectancy sub scale of the Credibility/Expectancy Questionnaire
Study safety | at the end of treatment at 6 weeks and 3 months after the end of treatment
  The proportion of participants that report no adverse events related to study participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD will be available from trial end through three years after the publication of all study results.
Access Criteria: Individuals will be able to access the data after signing a data sharing agreement.